CLINICAL TRIAL: NCT00189709
Title: A Single Center, Open, Parallel, Comparative, Randomized Study of Micafungin (FK463) vs Fluconazole (Diflucan) in the Treatment of Invasive Candidiasis and Candidaemia (Protocol No: MCFGCAN-0301F-TW)
Brief Title: Micafungin Versus Fluconazole in the Treatment of Invasive Candidiasis and Candidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCFGCAN-0301F-TW
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-01-02 (Estimated); Status verified 2007-12

CONDITIONS: Invasive Candidiasis; Candidemia
Keywords: micafungin; fluconazole; invasive candidiasis; candidemia
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia | interventions — Micafungin; Fluconazole

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Micafungin
- 2 (Active Comparator)
  Interventions: Drug: fluconazole

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: FK463
  Arms: 1
Drug: fluconazole — IV
  Other Names: Diflucan
  Arms: 2

SUMMARY:
To determine the efficacy and safety of micafungin (FK463) versus fluconazole (Diflucan) in treating patients with invasive candidiasis or candidaemia

DETAILED DESCRIPTION:
Micafungin (a new class of antifungal drugs) is compared to fluconazole (current standard treatment) in the treatment of patients with serious fungal infections (invasive candidiasis and candidemia) to determine its efficacy and safety. Patients, both male and female, aged over 16 and with confirmed disease by the doctor could be recruited and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of candidemia and invasive candidiasis
* Patients could be newly diagnosed with candidiasis who received no more than 48 hours of prior systemic antifungal therapy
* Inpatients aged 16 and above

Exclusion Criteria:

* Patients with serious invasive candidiasis whose prognoses are considered to be poor (life expectancy judged to be less than 5 days).
* Patients with severe complications in the liver
* Pregnant or lactating women
* Patients who have received at least 5 days of prior systemic treatment of fluconazole or echinocandin with no response.
* Patients who have prior antifungal infection requiring treatment with systemic antifungal agents for conditions other than candidemia and invasive candidiasis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Response rate | 2-8 Weeks

SECONDARY OUTCOMES:
Clinical response, mycological response | 2-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Chwen Chang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Taipei, Republic of China, Taiwan